CLINICAL TRIAL: NCT04491708
Title: What is the Metabolic Intensity of Pilates: An Analysis of the Energy Expenditure and Cardiovascular Markers of Intensity of Apparatus and Mat Pilates Sessions
Brief Title: What is the Metabolic Intensity of Pilates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Brasília (Other)
Responsible Party: Principal Investigator, Letícia de Souza Andrade, Clinical Professor, Catholic University of Brasília
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 28657514.0.0000.0029
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Energy Expenditure
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apparatus Pilates (Experimental): The same Pilates exercises were performed during the Mat Pilates and Reformer apparatus sessions. For each exercise, one set of 10 repetitions was performed. Between each exercise, participants were allowed to rest for 2 minutes in a lying position. For each exercise in the Reformer apparatus, the number of springs used was defined during the familiarization sessions as the highest number of springs the participant could perform the 10 repetitions of the exercise with proper technique and following the 5 Pilates principles correctly. The exercises performed were (Stott 2003; Stott 2001): 1) Cat stretch; 2) Hip rolls; 3) Ab prep; 4) Breast stroke preps; 5) Hundred; 6) Breast stroke; 7) Half roll back; 8) Single leg stretch; 9) Slow double leg stretch; 10) Double leg stretch; 11) Double leg circle; 12) Scissors; 13) Roll over; 14) Teaser; 15) Spine stretch forward.
  Interventions: Other: Pilates exercises
- Mat Pilates (Experimental): The same Pilates exercises were performed during the Mat Pilates and Reformer apparatus sessions. For each exercise, one set of 10 repetitions was performed. Between each exercise, participants were allowed to rest for 2 minutes in a lying position. For each exercise in the Reformer apparatus, the number of springs used was defined during the familiarization sessions as the highest number of springs the participant could perform the 10 repetitions of the exercise with proper technique and following the 5 Pilates principles correctly. The exercises performed were (Stott 2003; Stott 2001): 1) Cat stretch; 2) Hip rolls; 3) Ab prep; 4) Breast stroke preps; 5) Hundred; 6) Breast stroke; 7) Half roll back; 8) Single leg stretch; 9) Slow double leg stretch; 10) Double leg stretch; 11) Double leg circle; 12) Scissors; 13) Roll over; 14) Teaser; 15) Spine stretch forward.
  Interventions: Other: Pilates exercises

INTERVENTIONS:
Other: Pilates exercises — The participants attended two half-hour Pilates exercise classes twice a week, for one month, to familiarize themselves with the exercises and to learn the 5 Pilates' principles. After the learning period, two experimental sessions were performed: a Mat Pilates session and a Reformer apparatus Pilates session. The order of each session was randomized and drawn beforehand. Each experimental session lasted about one and a half hours and the interval between the sessions was 48 hours. Participants were asked to not perform any exercise and to refrain from food or fluids except water eight hours prior to each experimental session. Prior to the start of the experimental sessions, participants received a standard breakfast of 321 kcal that was 76% (61 g) carbohydrate, 8% (6,7 g) protein, 16% (5,9) fat, provided by the study researchers. All sessions were conducted at the same time in the morning, and the room temperature (22°C) and humidity (40-50%) were controlled during the whole session.

SUMMARY:
Background: Pilates is a form of structured physical activity that is commonly used in rehabilitation settings and to improve muscular fitness, balance, and flexibility. Despite its popularity, it is not known whether the energy expenditure (EE) and oxygen consumption from Pilates sessions could also lead to metabolic fitness benefits. The aim of this study was to quantify the intensity and the EE during two different types of Pilates sessions (mat and apparatus). Methods: 18 healthy females (age: 22 ± 3 years; height: 1.6 ± 0.1cm; body mass: 61.0 ± 10.0 kg; body mass index: 21 ± 3 kg/cm2) performed two different sessions. Each session involved the performance of 15 different exercises. Oxygen consumption (VO2) was measured continuously and then converted to EE in Kcal/min. Blood lactate, heart rate (HR), and blood pressure (BP) were also measured. A repeated measures two-way ANOVA (time X group) determined differences between types.

DETAILED DESCRIPTION:
The participants attended two half-hour Pilates exercise classes twice a week, for one month, to familiarize themselves with the exercises and to learn the 5 Pilates' principles. After the learning period, two experimental sessions were performed: a Mat Pilates session and a Reformer apparatus Pilates session. The order of each session was randomized and drawn beforehand. Each experimental session lasted about one and a half hours and the interval between the sessions was 48 hours. Participants were asked to not perform any exercise and to refrain from food or fluids except water eight hours prior to each experimental session. Prior to the start of the experimental sessions, participants received a standard breakfast of 321 kcal that was 76% (61 g) carbohydrate, 8% (6,7 g) protein, 16% (5,9) fat, provided by the study researchers. All sessions were conducted at the same time in the morning, and the room temperature (22°C) and humidity (40-50%) were controlled during the whole session.

Prior to the start of experimental sessions, participants rested in a supine position for 15 minutes. At the end of the 15 minutes, while still supine, measurements of BP and resting blood lactate were taken using standard laboratory procedures. Participants were then outfitted with a oxygen gas analyzer (Metalyzer 3b Cortex, Germany). Participants were connected by a mask, covering mouth and nose, to a digital gas flow analyzer. Standard calibration before every session was conducted according to the manufacturer's instructions.VO2 and HR were then simultaneously recorded for 5 minutes in a sitting position. At the end of the 5 minutes, the exercise session was started. VO2 and HR were monitored continuously throughout the session, while BP was assessed during rest intervals between exercises. At the end of the exercise session, BP and blood lactate were measured one time in a supine position in the post recovery time period. VO2 and HR were measured continuously for 5 minutes post session in a sitting position.

ELIGIBILITY:
Inclusion Criteria:

* Women aged up to 30 years;
* Sedentary or irregularly active, as assessed by the International Physical Activity Questionnaire (IPAQ);
* Not have any prior experience in Pilates exercises.

Exclusion Criteria:

* Have any clinical or orthopedic conditions/disease;
* Practitioner of any type of exercise.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | 50 minutes
  VO2 was measured continuously for both Mat and Reformer apparatus Pilates as described previously. Data were calculated on breath-by-breath intervals at rest and during exercise. The absolute EE in kilocalories per minute was estimated using a constant value of 5.05 kcal.L-1 O2, so the O2 values expressed in L/min were multiplied by 5.05. VO2 values in ml/min/kg were also considered for the analysis.

SECONDARY OUTCOMES:
Blood Lactate | 10 minutes
  Capillary blood samples were collected from a fingertip before the first exercise and immediately after the last exercise of the Mat Pilates and Reformer apparatus experimental sessions. These samples were added into a 3mL eppendorf tube with sodium fluorite and this mixture was frozen to be further analyzed via spectrophotometry using a YSI 2300 STAT Plus (Yellow Springs Instrument, Yellow Springs, Ohio, USA).
Heart rate | 50 minutes
  HR was recorded continuously throughout the sessions using a POLAR RS800cx heart-rate monitor (Polar Electro, Kempele, Finland) as per manufacturers guidelines for sensor belt placement. The mean HR of each Pilates sessions was determined using the Polar Precision Performance software (version 5.40.172).
Blood pressure | 15 minutes
  BP was measured using a digital BP monitor (Microlife BP 3BTO-A, São Paulo, Brazil) on the left arm. BP was measured, when participants lied on a bed on supine position, before, during (in the rest intervals between exercises) and after the exercises in the post exercise. Both pressures, sistolic and diastolic, was assessed during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yomara Mota, Study Director — Catholic University of Brasilia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilmore JH, Parr RB, Ward P, Vodak PA, Barstow TJ, Pipes TV, Grimditch G, Leslie P. Energy cost of circuit weight training. Med Sci Sports. 1978 Summer;10(2):75-8. PMID 692305